CLINICAL TRIAL: NCT01501435
Title: A Randomized, Open Label, Three-Treatment, Three-Period, Six-Sequence Crossover Study to Compare the Pharmacokinetics of CJ-30039 and Lipidil Supra and to Investigate Food-effect on Pharmacokinetics of CJ-30039
Brief Title: To Compare Safety and Pharmacokinetic Properties of CJ-30039 and Lipidil Supra
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CJ_FEN_101
Record Dates: First submitted 2011-12-24; First posted 2011-12-29 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Healthy
Keywords: Safety; Pharmacokinetics
MeSH Terms: interventions — fenofibric acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CJ-30039 (Experimental): Incrementally Modified Drugs of fenofibric acid
  Interventions: Drug: CJ-30039
- fenofibric acid (Active Comparator): Greencross Lipidil Supra 160mg
  Interventions: Drug: fenofibric acid

INTERVENTIONS:
Drug: CJ-30039 — single dose
  Other Names: Incrementally Modified Drugs of fenofibric acid
  Arms: CJ-30039
Drug: fenofibric acid — single dose
  Other Names: Greencross Lipidil Supra 160mg
  Arms: fenofibric acid

SUMMARY:
To investigate the safety and pharmacokinetic properties of CJ-30039 and Lipidil Supra

DETAILED DESCRIPTION:
Study objectives

* To compare the safety and pharmacokinetic properties of CJ-30039 and Lipidil Supra after a single oral administration in healthy male volunteers.
* To evaluate the food-effect on pharmacokinetics of CJ-30039 after a single oral administration in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male volunteers in the age between 20 and 55 years old
* BMI(Body Mass Index) in the range of 18.5 to 25kg/m2
* Subject with no history of any significant chronic disease

Exclusion Criteria:

* History of clinically significant allergies, including fenofibric acid or Fenofibrate
* History of clinically significant hepatic, renal, neurology, psychiatric, pulmonary, endocrine, hematologic, cardiovascular disease
* History of surgery except or gastrointestinal disease which might significantly change absorption of medicines
* Clinical laboratory test values are outside the accepted normal range

  * AST(ASpartate Transaminase), ALT(ALanine Transaminase)( > 1.25 times to normal range
  * Total bilirubin > 1.5 times to normal range
  * BUN(Blood Urea Nitrogen) > 25 mg/dL or Creatinine > 1.4 mg/dL
  * CK(Creatine Kinase) > 1.25 times to normal range
* Estimated GFR(Glomerular Filtration Rate) < 80 mL/min/1.73m2
* Clinically significant vital sign

  * SBP(Systolic Blood Pressure) ≤ 90 mmHg or SBP ≥ 150 mmHg
  * DBP(Diastolic Blood Pressure) ≤ 50 mmHg or DBP ≥ 100 mmHg
* History of drug abuse or positive urine screen for drugs
* History of caffeine, alcohol, smoking abuse

  * caffeine > 5 cups/day
  * alcohol > 201g/week
  * smoking > 10 cigarettes/day
* Use of prescription only medicine and oriental medicine within the 14 days before dosing or use of non-prescription medicine within the 7 days before dosing
* Participated in a previous clinical trial within 60 days prior to dosing
* Donated blood within 60 days prior to dosing

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2011-12; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of fenofibric acid | up to 48 hours

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of fenofibric acid | up to 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Min-su Park, MD PhD, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei university severance hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No